CLINICAL TRIAL: NCT07017101
Title: Effect of Neurophysiological Facilitation Techniques Applied in Addition to Pilates-based Exercise Training in Individuals With Fibromyalgia on Respiratory Parameters, Fatigue and Quality of Life
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Aliye Rabia AKKAYA, Effect of neurophysiological facilitation techniques applied in addition to pilates-based exercise training in individuals with fibromyalgia on respiratory parameters, fatigue and quality of life, Okan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: OKANU-FTR-ARA-01
Record Dates: First submitted 2025-05-19; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia (FM)
MeSH Terms: conditions — Fibromyalgia | interventions — Quality of Life

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PILATES BASED EXERCISE TRAINING WITH REFORMER (Experimental): Pilates training with reformer for 6 weeks
  Interventions: Other: PILATES BASED EXERCISE TRAINING WITH REFORMER
- NEUROPHYSIOLOGICAL FASCILITATION TECHNIQUES (Active Comparator): Control group
  Interventions: Other: PILATES BASED EXERCISE TRAINING WITH REFORMER; Other: NEUROPHYSIOLOGICAL FASCILITATION TECHNIQUES

INTERVENTIONS:
Other: PILATES BASED EXERCISE TRAINING WITH REFORMER — Participants will only be given training on pilates-based exercises with reformers. Breathing, which are the 5 key elements of clinical pilates exercises after the first evaluation to individuals,
  Focus, rib cage placement, shoulder placement, head and neck placement will be taught. Whole
  Participants will be informed about the reformer instrument and work schedule. Exercises 2 days a week, 6
  Will be applied throughout the week.
  Other Names: Effect of neurophysiological facilitation techniques applied in addition to pilates-based exercise training in individuals with fibromyalgia on respiratory parameters, fatigue and quality of life
Other: NEUROPHYSIOLOGICAL FASCILITATION TECHNIQUES — In addition to reformer-based pilates training, participants will be given Neurophysiological facilitation techniques training. Neurophysiological facilitation techniques are non-invasive, easy to apply, the physiotherapist is active
  It consists of exercises made with guidance and active participation of the patient. These techniques are any
  Does not contain an electrotherapy current. In this study, the neurophysiological
  Facilitation techniques, perioral stimulation, intercostal tension, anterior basal lift, vertebral pressure, medium
  Graded manual pressure and abdominal co-contraction techniques and each technique for 15 seconds
  Will be applied. Neurophysiological facilitation techniques are used to repeat 10 sessions each session throughout the treatment.
  It will be done.
  Other Names: Effect of neurophysiological facilitation techniques applied in addition to pilates-based exercise training in individuals with fibromyalgia on respiratory parameters, fatigue and quality of life
  Arms: NEUROPHYSIOLOGICAL FASCILITATION TECHNIQUES

SUMMARY:
The aim of our study was to examine the effect of neurophysiological facilitation techniques applied in addition to pilates-based exercise training in individuals with fibromyalgia on body composition, core stabilization, respiratory parameters, fatigue and quality of life.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic musculoskeletal problem characterized by widespread pain in the body accompanied by other symptoms such as fatigue, sleep disturbance, morning stiffness and increased sensitivity in some anatomical areas. Chronic pain in FM causes physical and emotional stress and can reduce quality of life. In FM management, it is recommended to combine pharmacological and non-pharmacological methods with the active participation of the person. Exercise is an important part of non-pharmacological approaches. The purpose of exercise in FM management is to reduce pain and fatigue, increase muscle strength, flexibility and endurance, and contribute to the person's functionality, quality of life. Exercise also provides relaxation and causes healing effects in the emotional state. Recent studies have shown that the use of clinical pilates exercises has become popular in individuals with fibromyalgia.

Pilates was developed by Joseph Humbertus Pilates in the early 1900s and was adapted by health professionals for therapeutic use and called "Clinical Pilates". It is a popular exercise method used in both healthy and patient populations today. Clinical Pilates exercises train the mind to consciously focus on controlling the movement and posture of the body. It aims to improve the relationship between mind and body with the active participation of the patient. It is also different from other types of exercise because it contains a breathing component. Pilates exercises can be applied in two methods: mat pilates and equipment pilates. Mat pilates exercises are done on a mat, while equipment pilates exercises are done using special types of equipment such as reformer, cadillac, wunda chair, ladder barrel.

Reformer is the most popular equipment among pilates equipment. It consists of springs, rollers, ropes and a sliding platform that provide variable resistance. Joseph Pilates believed that starting exercise in a moving/sliding horizontal plane and advancing other exercises with additional gravitational forces added was important to reduce stress on the joints. Therefore, he designed the reformer that allowed the exercises to be applied to the horizontal plane. Exercises with the reformer are done against resistance in the horizontal plane, where gravity is eliminated. Reformer exercises focus on maintaining the neutral position and quality of body alignment, and also exercises can be done in different positions, such as kneeling, lying on the side, standing. Some studies show that pilates exercises applied with reformer, pain and balance in working women with chronic low back pain (Basakcı Calık et al., 2018), pain, function and kinesophobia in individuals with chronic low back pain (Altan et al. 2009 - Patti et al., 2015) has shown positive effects on balance, functionality, cor stabilization, fatigue severity and quality of life in patients with multiple sclerosis (Frank et al., 2017).Although mat pilates has been shown to be an effective and safe treatment method to reduce symptoms in individuals with fibromyalgia, studies for the effects of reformer pilates in FM are limited (Korkmaz, 2010- Palekar, 2014). The literature has shown that mat pilates exercises for individuals with FM are usually performed as a supervised schedule (Franco et al., 2019). Neurophysiological facilitation techniques are a non-invasive exercise technique and are based on the combination of maximal resistance applied during the joint range of motion with posture and stretching reflexes and primitive movement patterns (Çetintaş and Kamanlı, 2012). Hand contacts, communication with the patient, stretching, traction, aproximation, maximal resistance applications, strengthening methods, facilitation techniques applied to ensure harmonious and indequent contractions of the muscles (Çetintaş and Kamanlı, 2012). These exercises do not include any electrotherapy methods. It is an exercise approach aimed at improving movement and function using the natural working principles of the nervous system and muscles. In this method, movement patterns are used that allow the muscles to work together and coordinate the movement of the nervous system (Çetintaş and Kamanlı, 2012). Proprioceptive Neuromuscular Fascitation (PNF) is defined as facilitating the responses of the neuromuscular mechanism by stimulation of proprioceptors. The basic principle of PNF is based on the fact that the movements in the human body have a rotational and oblic character and a greater response can be obtained with the movement against maximum resistance. PNF exercises are useful for pain in individuals with fibromyalgia. At the same time, the sensory-motor system is effective in regulation and balance development. Rhythmic stabilization technique and Pilates motor control exercises have been shown to lead to significant improvement in pain and joint range of motion (Malla, 2018). In a study comparing PNF exercises and the McKenzie method in individuals with fibromyalgia, the combined isotonic contraction technique with the PNF rhythmic stabilization technique was shown to be effective in improving the quality of life of individuals (Anggiat et al., 2018). In another study in individuals with fibromyalgia, the PNF combined isotonic contraction technique was shown to provide the benefit of improving functional capacity and reducing pain (Zaworski and Latosiewicz, 2018). It is stated that PNF exercises contribute to reducing pain, increasing muscle strength and functional capacity and quality of life (Arslan and Erbahçeci, 2016). In studies using pilates exercises and PNF exercises in the literature, both methods have been shown to have an effect on some parameters such as fibromyalgia pain, functional level and quality of life. Studies in the literature show that both methods are among the treatment methods frequently used in the clinic by physiotherapists, but it is difficult to provide adequate information about which method is more effective. In the light of this information, the aim of our study is to examine the effect of neurophysiological facilitation techniques applied in addition to pilates-based exercise training in individuals with fibromyalgia on body composition, cor stabilization, respiratory parameters, fatigue and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Being between the ages of 18-65,

Having been diagnosed with FM by a specialist physician according to ACR 2016 criteria

Volunteering to participate in the study,

Exclusion Criteria:

Not showing voluntary participation in the study,

Orthopedic, neurological and cardiopulmonary diseases that will prevent him from exercising

Existence,

Pregnancy,

Having exercised regularly for the last 3 months,

Individuals with a known history of psychiatric illness and receiving active psychiatric treatment

Will be excluded from research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-06-21 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Effect of neurophysiological facilitation techniques applied in addition to pilates-based exercise training on respiratory parameters, fatigue and quality of life in individuals with fibromyalgia | 6 weeks after registration

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Aydın, Study Director — Okan Üniversitesi
Locations (1):
- RA Fizyoterapi, Istanbul, Tuzla, Turkey (Türkiye)